CLINICAL TRIAL: NCT05940987
Title: Phone-based Smoking Cessation Intervention for Patients With Chronic Pancreatitis ：a Prospective Multicenter Randomized Clinical Trial
Brief Title: Phone-based Smoking Cessation Intervention for Patients With Chronic Pancreatitis.(START)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, professor, Changhai Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: START
Record Dates: First submitted 2023-06-15; First posted 2023-07-12 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Pancreatitis, Chronic
Keywords: Smoking Cessation; Phone-based intervention
MeSH Terms: conditions — Pancreatitis, Chronic; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): Participants in the intervention group will receive one 20-30 minutes "5A" smoking cessation health consultation after enrollment; They will be given regular phone-based smoking cessation intervention once a week in the first month and once a month thereafter (15 times in total). Participants will be followed at 2, 6, 12 months, and cotinine urine test kits will be mailed to those who have self-reported smoking cessation at follow-up, which is used to confirm whether they have quitted smoking or not. (smoking cessation is defined as urine cotinine levels below 200 ng/mL).
  Interventions: Behavioral: Phone-based smoking cessation intervention
- Control Group (No Intervention): Participants in the control group will receive one 20-30 minute "5A" smoking cessation health consultation after enrollment; Phone-based smoking cessation intervention will not be regularly given after enrollment.

INTERVENTIONS:
Behavioral: Phone-based smoking cessation intervention — Participants who allocate to the intervention group will receive regular phone-based smoking cessation intervention by professional team.
  Arms: Intervention Group

SUMMARY:
This study aims to explore whether regular telephone intervention in patients with chronic pancreatitis can improve their smoking cessation rate.

DETAILED DESCRIPTION:
Chronic pancreatitis（CP） is a chronically progressive disease characterized by pancreatic fibrosis and inflammation, and its basic pathological features include chronic inflammatory damage to the pancreatic parenchyma, interstitial fibrosis, pancreatic parenchymal calcification, pancreatic duct dilation, and pancreatic duct stones.

Environmental factors such as alcoholism，smoking and genetic factors are the main causative factors of CP. Clinical studies have found that smoking can not only accelerate the course of CP, but also increase the risk of CP-related complications. Some scholars believe that smoking cessation may be a potential way to prevent the progression of CP and improve the prognosis of CP. Although there is no evidence to verify whether smoking cessation will improve the clinical course of CP, the latest ACG Clinical Guideline strongly recommends CP patients quit smoking.

In 2016，a prospective study of smoking cessation interventions in CP patients showed that 27 enrolled patients had a smoking cessation rate of 0% after 6 months of smoking cessation intervention, indicating that smoking cessation is a huge challenge for CP patients.

The investigators propose to conduct a randomized controlled trial to investigate the effects of telephone intervention on smoking cessation in patients with CP and explore the impact of smoking cessation on their clinical course and prognosis.

ELIGIBILITY:
Inclusion Criteria:

1.18 years of age and older living; 2.Patients diagnosed as chronic pancreatitis; 3.Self-reported smoking ≥ 5 cigarettes; 4.Urine cotinine levels ≥ 200 ng/mL; 5.Owning a phone; 6.Willing to provide informed consent to participate in the study.

Exclusion Criteria:

1. Patients diagnosed as pancreatic cancer within 2 years after diagnosing chronic pancreatitis; Patients diagnosed as groove pancreatitis or autoimmune pancreatitis;
2. Pregnant or lactating women;
3. Patients with life expectancy ≤ 12 months;
4. Comorbidities such as Alzheimer's disease, end-stage cancer, HIV, end-stage congestive heart failure, end-stage chronic obstructive pulmonary disease, uncompensated cirrhosis, renal failure;
5. Smoking e-cigarettes or other forms of non-burning tobacco.
6. Patients refused to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 382 (Actual)
Dates: Start 2023-06-28 (Actual); Primary Completion 2025-02-25 (Actual); Study Completion 2025-02-25 (Actual)

PRIMARY OUTCOMES:
Biochemically Validated of 7-day Point Abstinence | 12 months
  The primary outcome will be biochemical validation of Self-reported 7-day point-prevalence abstinence at month 2, 6, 12 after quit date.

SECONDARY OUTCOMES:
Self-reported 7-day Point Abstinence | 12 months
  Self-reported 7-day point-prevalence abstinence at month 2, 6, 12 after quit date.
Number of cigarettes smoked per day | 12 months
  Mean number of cigarettes smoked per day among participants still smoking at 12 months.
Fagerstrom Test of Nicotine Dependence (FTND) scores | 12 months
  The FTND is a validated, 6-item self-report instrument that evaluates the intensity of physical addiction to nicotine. The scores will be assessed at month 2, 6, 12 after quit date.Three items are rated yes/no (0/1), and the other three items are rated on a scale from 0-3. Items are summed to yield a total score of 0-10, with higher scores reflecting greater nicotine dependence. This outcome variable will be reported as the difference in FTND total score between the intervention condition and the control condition.

OTHER OUTCOMES:
Reduction in Tobacco Consumption | 12 months
  The number of CP patients who self-reported a 50% reduction in tobacco consumption at 2, 6 and 12 months after quit date.
Times of hospitalizations | 12 months
  The times of hospitalizations for episodes of chronic pancreatitis at 12 months after quit date.

CONTACTS AND LOCATIONS:
Overall Officials: Liang-hao Hu, M.D., Principal Investigator — Changhai Hospital
Locations (1):
- Changhai Hostipal, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No